CLINICAL TRIAL: NCT02622217
Title: Impact of Sleep Deprivation on Anesthesiology Residents' Non-technical Skills: a Simulation Based Randomised Study.
Brief Title: Impact of Sleep Deprivation on Anesthesiology Residents' Non-technical Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Paris 5 - Rene Descartes (Other)
Responsible Party: Principal Investigator, Arthur Neuschwander, Dr, University of Paris 5 - Rene Descartes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UParis5
Record Dates: First submitted 2015-11-28; First posted 2015-12-04 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Sleep Deprivation
Keywords: anesthesiology; non technical kills
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep deprived (Experimental): Participants undergo a simulation session after an on call night
  Interventions: Behavioral: Sleep deprivation
- Rested (No Intervention): Participants undergo a simulation session after a night of normal sleep at home

INTERVENTIONS:
Behavioral: Sleep deprivation
  Arms: Sleep deprived

SUMMARY:
Sleep deprivation is common in anaesthesiology residents. Its effects on technical skills have been reported with controversial results. Non-technical skills (team working, situation awareness, decision making and task management) contribute to safe and efficient task performance. They have a crucial role in anaesthetic practice, especially during crisis management. The investigators hypothesized that sleep deprivation was associated with a reduced mobilisation of non-technical skills in anaesthesiology residents.

DETAILED DESCRIPTION:
The scenario consisted in a rapid sequence induction for emergency general anaesthesia in case of acute peritonitis complicated by an anaphylactic shock secondary to the injection of succinylcholine. All scenarios were performed with the assistance of an anaesthetist nurse, facilitator of the scenario. In a second time, after patient stabilisation (defined as oxygen saturation by pulse oximetry (SpO2) > 95%, mean arterial pressure (PAM) > 65 mmHg and heart rate (HR) < 100 bpm for at least 2 minutes) consecutive to an expected injection of 100 µg of epinephrine decided by the participant, a surgeon entered the operating room to create a dilemma regarding patient destination (continue surgery or intensive care unit admission)

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology residents from Paris academic hospitals

Exclusion Criteria:

* Chronic sleep disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Anesthetists non technical skills (ANTS) scale | day 0 during procedure
  score assessed by 2 blinded evaluators during scenario

SECONDARY OUTCOMES:
Technical skills | day 0 during procedure
  Check list of items, assessed by 2 blinded evaluators during scenario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Neuschwander A, Job A, Younes A, Mignon A, Delgoulet C, Cabon P, Mantz J, Tesniere A. Impact of sleep deprivation on anaesthesia residents' non-technical skills: a pilot simulation-based prospective randomized trial. Br J Anaesth. 2017 Jul 1;119(1):125-131. doi: 10.1093/bja/aex155. PMID 28974071